CLINICAL TRIAL: NCT01018524
Title: Results of Open Mesh Versus Suture Repair in Treatment of Abdominal Wall (Multicentric, Prospective, Randomised, Internet-based, Clinical Trial)
Brief Title: Open Mesh Versus Suture Repair in Treatment of Abdominal Wall Hernias
Acronym: HSS-AHS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hungarian Surgical Society (Network)
Responsible Party: Prof. Dr. O.P. Horvath, Hungarian Surgical Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HSS-AHS 02-09
Record Dates: First submitted 2009-10-13; First posted 2009-11-23 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Abdominal Hernia
Keywords: position of the mesh; recurrence rate; surgical procedure; long time outcome
MeSH Terms: conditions — Hernia, Abdominal | interventions — Abdominoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- small hernias - suture repair (Active Comparator)
  Interventions: Procedure: abdominal wall reconstruction
- small hernias - mesh repair (Active Comparator)
  Interventions: Procedure: abdominal wall reconstruction
- large hernias - sublay mesh (Active Comparator)
  Interventions: Procedure: abdominal wall reconstruction
- large hernias - onlay mesh (Active Comparator)
  Interventions: Procedure: abdominal wall reconstruction

INTERVENTIONS:
Procedure: abdominal wall reconstruction — suture repair, mesh repair, onlay mesh reconstruction, sublay mesh reconstruction, recurrence rate

SUMMARY:
The purpose of this study is to:

1. compare the long term results of mesh versus suture repair in treatment of abdominal wall defects;
2. find the optimal location of implanted prosthesis, comparing the two most useful position of mesh in abdominal wall hernia surgery.

DETAILED DESCRIPTION:
To determine difference of operation time, applied materials of hernia operations; clinical complications, postoperative pain, hernia recurrence, recovery and normal activity time after surgery.

ELIGIBILITY:
Inclusion Criteria:

* During the two-year randomization period at the joined centres all patients were included who were admitted with abdominal wall or umbilical hernia and who suited the requirements.
* All the patients with primer or first recurrence of postoperative abdominal or primer or first recurrence of umbilical hernia were randomized into this study.
* For involvement into the study good patient compliance, signed consent form, normal local circumstances were needed.

Exclusion Criteria:

* Ages fewer than 18 or above 70 years
* Hernia orifice under 5 cm2.
* Planned or accidental intraoperative opening of any bowel.
* Unstable parameters of circulation, uncontrollable diabetic or autoimmune disease.
* Severe renal or hepatic failure
* Advanced stage of tumours or currently treated malignancies.
* Inflamed or muddy content of hernia sac.
* If the patient did not signed the consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
recurrence rate after hernia surgery | 5 years

SECONDARY OUTCOMES:
chronic pain after hernia surgery | more one year
complications after hernia surgery | 0-5 years

CONTACTS AND LOCATIONS:
Overall Officials: György Wéber, Prof. Dr., Principal Investigator — Hungarian Surgical Society; József Baracs, Dr., Study Director — Hungarian Surgical Society
Locations (1):
- Dept. of Surgery Univ. of Pecs, Pécs, Hungary

REFERENCES:
- [Background] Weber G, Horvath OP. [Results of ventral hernia repair: comparison of suture repair with mesh implantation (onlay vs sublay) using open and laparoscopic approach--prospective, randomized, multicenter study]. Magy Seb. 2002 Oct;55(5):285-9. Hungarian. PMID 12474512
- [Derived] Weber G, Baracs J, Horvath OP. ["Onlay" mesh provides significantly better results than "sublay" reconstruction. Prospective randomized multicenter study of abdominal wall reconstruction with sutures only, or with surgical mesh--results of a five-years follow-up]. Magy Seb. 2010 Oct;63(5):302-11. doi: 10.1556/MaSeb.63.2010.5.3. Hungarian. PMID 20965863